CLINICAL TRIAL: NCT02329951
Title: Prospective, Observational Study Evaluating the Ability of Clinical Factors to Predict Interventional Treatment Outcomes for Low Back Pain (LBP)
Brief Title: Predictive Factors for LBP Interventional Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Landstuhl Regional Medical Center (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB00050132
Record Dates: First submitted 2014-12-30; First posted 2015-01-01 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain; Lumbar Radiculopathy
MeSH Terms: conditions — Low Back Pain; Radiculopathy | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Epidural steroid injections: Patients will receive a single interlaminar epidural steroid injection with 60 mg depomethylprednisolone, 1.5 ml of 0.25% bupivacaine and 1.5 ml of saline or a transforaminal epidural steroid injection with 60 mg depomethylprednisolone, 1.5 ml of 0.25% bupivacaine and 0.5 ml of saline.
  Interventions: Procedure: Epidural steroid injection
- Facet interventions: Patients will receive diagnostic medial branch (facet joint nerve) blocks with 0.5 ml of 0.5% bupivacaine. If they experience a positive block (> 50% pain relief lasting more than 3 hours), they will then receive radiofrequency denervation.
  Interventions: Procedure: Facet intervention
- Sacroiliac joint injections: Patients will receive a single SI joint injection on the affected side(s) with 40 mg depomethylprednisolone and 2 ml of 0.5% bupivacaine.
  Interventions: Procedure: Sacroiliac joint injection

INTERVENTIONS:
Procedure: Facet intervention — Diagnostic block of the nerves innervation the lumbar facet joint. If this block is positive (greater or equal to 50% relief), the participant will proceed to radiofrequency nerve ablation when the pain returns
  Other Names: Medial branch block and radiofrequency ablation
  Groups: Facet interventions
Procedure: Sacroiliac joint injection — Injection of steroid and local anesthetic into SI joint
  Groups: Sacroiliac joint injections
Procedure: Epidural steroid injection — Transforaminal or interlaminar injection of steroid epidurally
  Groups: Epidural steroid injections

SUMMARY:
In this study, we are attempting to determine which factors are associated with interventional treatment outcome for LBP (and to what extent). Up to 346 patients with LBP who are considered to be good candidates for therapeutic interventional procedures will be given a complete history and physical exam, which includes the assessment of Waddell signs, and querying them regarding factors shown in non-interventional studies or retrospective studies evaluating interventional treatments to be associated with negative treatment outcomes. These factors include the presence of Waddell and other physical exam signs, opioid use, allergies, psychopathology, concomitant pain conditions, a 6-point Likert scale on expectations, sleep abnormalities, secondary gain (e.g. medical board or litigation), procedure-related pain including from a 1 ml standardized injection, obesity, and smoking history. They will then proceed to undergo their scheduled intervention, which will be limited to epidural steroid injections (ESI), facet blocks and if positive, radiofrequency denervation, and sacroiliac (SI) joint injections. A positive outcome will be defined as 2-point or greater decrease in average pain score at 1-month and a score of > 3 on a 1-5 Likert satisfaction scale. Those with a positive outcome at 1-month will remain in the study and be followed again at 3-months.

DETAILED DESCRIPTION:
This will be an observational study with a 3-month follow-up. The course of clinical treatment will be decided by a physician independent of the research. Besides filling out questionnaires and standardized follow-up visits, all subjects will receive the same care they would if they did not participate in the study. The study will be discussed with the subjects and they will be enrolled in the study after it is determined that they meet selection criteria and are scheduled for one of the above injections. They will then fill out 3 questionnaires (Oswestery disability index, Athens insomnia scale, QIDS SR-16. All procedures will be performed with fluoroscopy. Following each procedure, the procedure-related pain will be reported on a 0-10 scale (all patients will receive as much 1% lidocaine local anesthetic as is necessary), including the reported pain to the standardized skin wheal at the start of the procedure.

Patients will then receive standardized epidural steroid injections (transforaminal or interlaminar), sacroiliac joint injections, or facet blocks and radiofrequency denervation if they experience a positive block. Details about these procedures are available upon request.

No patients will be permitted additional interventions between the time of their procedure and follow-up visits. Rescue medications will be in the form of either tramadol, NSAIDs or if the patient is on opioids, a < 20% increase in dose. The first follow-up visit will be scheduled 1 month from the start of treatment for ESI and SI joint patients, and 1 month after RF denervation in positive diagnostic facet block responders. In those facet block patients who obtain prolonged relief from the "diagnostic" medial branch block, follow-up will be 1 month after the block (these patients may proceed to have denervation if their pain recurs after 1 month but before their final 3-month follow-up, and their 3-month follow-up will be 3 months after their medial branch block). A positive outcome will be defined as a greater or equal to 2-point decrease in average LBP (or leg pain for those who underwent an ESI) coupled with a positive satisfaction rating (> 3 on a 5-point scale). Subjects who obtain a positive outcome at their initial 1-month follow-up visit will remain in the study and return for the final 3-month follow-up visit. Those with a negative outcome will exit the study "per protocol" to receive standard care, which may consist of other injections or non-rescue medications such as antidepressants and anticonvulsants. Subjects who obtain a positive outcome at 1-month but experience a recurrence before their 3-month follow-up visit will also exit the study per protocol, with their final outcome measures recorded before they receive standard care.

In those who receive ESI, a smaller parallel study will be done evaluating the association between allergies and outcome. Allergies will be categorized as immunologically based or not.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Pain duration > 6 weeks;
3. Low back pain presumed to be secondary to herniated disc or spinal stenosis (e.g. radiculopathy), facet joint pain or SI joint pain;
4. For ESI, patients must have leg pain >/= 4/10 or comparable or greater than back pain, along with concordant MRI findings; for SI joint injections, patients must have tenderness overlying the SI joint; for facet joint pain, they must have paraspinal tenderness;
5. Patient agrees to have ESI, facet blocks or SI joint injection for diagnostic or therapeutic purposes;
6. Average pain score >/= 4/10 over the past week

Exclusion Criteria:

1. Previous ESI, facet blocks or SI joint injection within the past 2 years;
2. Active inflammatory spondyloarthropathy (e.g. ankylosing spondylitis);
3. Previous surgery for ESI or facet block;
4. Untreated coagulopathy;
5. Allergy to contrast dye, bupivacaine or depomethylprednisolone;
6. Pregnancy;
7. Cannot read or understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with low back or lumbar radicular pain scheduled for an injection
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Mean reduction in average pain score | 1 month
  0-10 numerical rating scale for leg pain (ESI) or low back pain (facet procedure or sacroiliac joint injection). Higher scores indicate more pain.

SECONDARY OUTCOMES:
Average back pain score | 1 month
  0-10 numerical rating scale for back pain. Higher scores indicate more pain.
Average leg pain score | 1 month
  0-10 numerical rating scale for leg pain for ESI only. Higher scores indicate more pain.
Worst back pain score | 3 months
  0-10 numerical rating scale for back pain. Higher scores indicate more pain.
Worst leg pain score | 3 months
  0-10 numerical rating scale for leg pain ESI only. Higher scores indicate more pain.
Oswestry disability index score | 1 month
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Oswestry disability index score | 3 months
  0-100% score measuring function for back and/ leg pain (higher scores indicate worse function)
Satisfaction score | 1 month
  5-point Likert scale measuring satisfaction (higher scores indicate greater satisfaction)
Satisfaction score | 3 months
  5-point Likert scale measuring satisfaction (higher scores indicate greater satisfaction)
Medication reduction | 1 month
  Cessation of non-opioid analgesic or > 20% change in opioids (yes or no)
Medication reduction | 3 months
  Cessation of non-opioid analgesic or > 20% change in opioids (yes or no)
Athens Insomnia Scale | 1 month
  0-24 point scale measuring sleep quality (higher scores indicate greater sleep dysfunction)
Athens Insomnia Scale | 3 months
  0-24 point scale measuring sleep quality (higher scores indicate greater sleep dysfunction)
Quick Inventory of Depressive Symptomatology (QIDS-SR 16) | 1 month
  0-48 point scale measuring symptoms of depression (higher scores indicate greater depressive symptoms)
Quick Inventory of Depressive Symptomatology (QIDS-SR 16) | 3 months
  0-48 point scale measuring symptoms of depression (higher scores indicate greater depressive symptoms)
Positive outcome | 1 month
  Greater or equal to 2-point change in back pain (facet procedure or sacroiliac joint injection) or leg pain (ESI) plus > 3 score on the 1-5 satisfaction scale. This is either yes or no.
Positive outcome | 3 months
  Greater or equal to 2-point change in back pain (facet procedure or sacroiliac joint injection) or leg pain (ESI) plus > 3 score on the 1-5 satisfaction scale. This is either yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Cohen SP, Doshi TL, Kurihara C, Reece D, Dolomisiewicz E, Phillips CR, Dawson T, Jamison D, Young R, Pasquina PF. Multicenter study evaluating factors associated with treatment outcome for low back pain injections. Reg Anesth Pain Med. 2022 Feb;47(2):89-99. doi: 10.1136/rapm-2021-103247. Epub 2021 Dec 8. PMID 34880117
- [Derived] Cohen SP, Doshi TL, Kurihara C, Dolomisiewicz E, Liu RC, Dawson TC, Hager N, Durbhakula S, Verdun AV, Hodgson JA, Pasquina PF. Waddell (Nonorganic) Signs and Their Association With Interventional Treatment Outcomes for Low Back Pain. Anesth Analg. 2021 Mar 1;132(3):639-651. doi: 10.1213/ANE.0000000000005054. PMID 32701541